CLINICAL TRIAL: NCT03409146
Title: Accuracy and Reliability of a New Intrapartum Fetal Heart Rate, Maternal Heart Rate, and Uterine Contraction Monitoring Method Compared With Food and Drug Administration (FDA) Approved Techniques.
Brief Title: Accuracy and Reliability of Novii: Fetal Heart Rate (FHR), Maternal Heart Rate (MHR) and Uterine Contraction (UA) Compared With Doppler, Scalp Fetal Scalp Electrode (FSE), Tocodynamometer (TOCO) and Intra Uterine Pressure Catheter (IUPC)
Status: Completed | Type: Observational
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 1404298207
Record Dates: First submitted 2018-01-11; First posted 2018-01-24 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Term Labour

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Term Patients: Approximately 80 pregnant women monitored in labor between 37 and 42 weeks' gestation will be necessary to complete the study. Subjects will have a singleton >37 week pregnancy.
  Subjects will be recruited for the study in the following groups :
  At least 10 patients with Body Mass Index (BMI) < 30 kg/m2 At least 10 patients with BMI 30-34.9 kg/m2 At least 10 patients with BMI ≥ 35 kg/m2
  Interventions: Device: Monica Novii Wireless Patch System

INTERVENTIONS:
Device: Monica Novii Wireless Patch System — The Monica Novii Wireless Patch System is a transabdominal fetal/maternal recorder that provides fetal heart rate, maternal heart rate and maternal uterine activity contractions.

SUMMARY:
Accuracy and Reliability of the Novii device (fetal heart rate, maternal heart rate and uterine activity) compared with Food and Drug Administration (FDA) approved techniques

DETAILED DESCRIPTION:
The study is being done to test the performance of a Novii Wireless Patch System for following the baby's and mother's heart rates and uterine contractions during labor. We want to find out if the new monitor works as well as other types of monitors that are usually used: Doppler Fetal Heart Rate (FHR), Scalp FHR, Tocodynamometer (TOCO) and Intra Uterine Pressure Catheter (IUPC).

80 patients will be monitored during the study.

ELIGIBILITY:
Inclusion Criteria:

A woman will be considered for inclusion in the study if she fulfills all of the following criteria:

* She has a term or near term (≥36 completed weeks) singleton gestation in a cephalic presentation and has been admitted to the Labor and Delivery Unit .
* She is in the latent phase of spontaneous labor, or has been admitted for induction of labor.
* She has given her informed consent to participate as a subject.
* She has none of the exclusion criteria.

Exclusion Criteria:

* Known major fetal malformation or chromosome abnormality.
* Multiple gestation
* A condition for which cesarean will likely be carried out shortly.
* Subject plans not to have electronic fetal monitoring.
* Involvement in another clinical trial currently or previously in this pregnancy that, in the investigator's opinion, would affect the conduct of this study.
* Medical or obstetric problem that would preclude the use of abdominal electrodes (e.g., skin eruptions, history of sensitivity to adhesives).
* Parturient is under age 18.
* Medical or obstetric problem that in investigator's opinion would make the patient incapable of taking part in the study.
* Inability to understand the consent information due to medical illness or diminished intellectual capacity, or insurmountable language barrier.
* Potential for coercion, e.g. Medical Center employees, prisoners.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women at term
Study Population: Pregnant Women at Term
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-05-28 (Actual); Primary Completion 2017-02-13 (Actual); Study Completion 2017-02-13 (Actual)

PRIMARY OUTCOMES:
Fetal Heart Rate (FHR) Positive Percentage Agreement (PPA) | through study completion, an average of 1 year
  PPA(%)=(a/(a+C))x100, where "a" represents the number of 2 second epochs when the Novii FHR is within +/-10% of the predicate device FHR for each 2 second epoch, and "c" are the number of 2 second epochs when the Novii FHR is not within +/- 10% of the predicate device FHR or is absent.

SECONDARY OUTCOMES:
Mean Percentage FHR Equivalence | through study completion, an average of 1 year
  The 2 second output FHR data when both the predicate and Novii devices are reporting a value will be considered. In this case for each 2 second epoch the FHR value from the Novii device is divided by the predicate device FHR value to create a "FHR ratio".
Uterine Activity (UA) Sensitivity (from Individual Contractions) | through study completion, an average of 1 year
  The Sensitivity of the Novii System against the predicate device is determined from the "individual contraction "detection as follows: Sensitivity(%)=(x/(x+z))x100
  Where:
  "x" is the total number of "individual contractions" detected by both the devices "z" is the total number of "individual contractions" detected by the predicate device only
Uterine activity Positive Percentage Agreement (from Interpretable Data) | through study completion, an average of 1 year
  The positive percentage agreement (PPA) is determined from the interpretable and uninterpretable data as follows:
  PPA(%)=(a/(a+c))x100
  Where:
  "a" is the number of minutes when both devices UA are "interpretable" at the same time "c" is the number of minutes when the predicate device UA is "interpretable" but the Novii system UA is "un-interpretable".
Maternal Heart Rate (MHR) Positive Percentage Agreement (PPA) | through study completion, an average of 1 year
  PPA(%)=(a/(a+C))x100, where "a" represents the number of 2 second epochs when the Novii MHR is within +/-10% of the predicate device MHR for each 2 second epoch, and "c" are the number of 2 second epochs when the Novii MHR is not within +/- 10% of the predicate device MHR or is absent.
Mean Percentage MHR Equivalence | through study completion, an average of 1 year
  The 2 second output MHR data when both the predicate and Novii devices are reporting a value will be considered. In this case for each 2 second epoch the MHR value from the Novii device is divided by the predicate device MHR value to create a "MHR ratio".

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona Medical Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No